CLINICAL TRIAL: NCT00133484
Title: A Phase II Study to Assess the Safety, Tolerability, Immunogenicity, and Optimal Primary Schedule of 3 Recombinant Protective Antigen (rPA) Anthrax Vaccines Administered in Two Intramuscular Doses to Healthy Adults
Brief Title: UMD rPA Regimen Trial in Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-026; Anthrax CVD 3000
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-12

CONDITIONS: Bacillus Anthracis (Anthrax)
Keywords: Anthrax, rPA
MeSH Terms: conditions — Anthrax | interventions — Replication Protein A

INTERVENTIONS:
Biological: Anthrax vaccine absorbed made from Bacillus anthracis (AVA)
Biological: Recombinant protein antigen (rPA) made from Bacillus anthrax
Biological: Recombinant protein antigen (rPA) made from Escherichia coli

SUMMARY:
Objectives are: To confirm the safety and tolerability of 2-dose regimens of 100 g rPA vaccines (3 products) administered by the intramuscular (IM) route to healthy adults.To describe the immunologic responses to 2-dose regimens of 3 rPA vaccines and to compare the responses to those following administration of Anthrax Vaccine Adsorbed (AVA or BioThraxTM), the currently available vaccine. The primary immunologic outcome is the proportion of volunteers in each group that mounts an antibody response (defined as a 4-fold or greater increase from pre-vaccination to post-vaccination of anti-rPA IgG antibody with a minimal concentration of 10 µg/ml as measured by ELISA). Secondary outcomes are time to peak response and GMC of anti-PA antibody at peak for each group. In addition, the following immunologic assays will be performed: toxin neutralization assay, oral fluid ELISA, antibody avidity, IgG subclasses, and B-cell memory,T-cell memory and effector subpopulations.

DETAILED DESCRIPTION:
Anthrax CVD 3000: A Phase II Study to Assess the Safety, Tolerability, Immunogenicity, and Optimal Primary Schedule of 3 Recombinant Protective Antigen (rPA) Anthrax Vaccines Administered in Two Intramuscular Doses to Healthy Adults aged 18 to 50 years. The targeted number of subjects is 270.The study objectives are:To confirm the safety and tolerability of 2-dose regimens of 100 g rPA vaccines (3 products) administered by the intramuscular (IM) route to healthy adultsTo describe the immunologic responses to 2-dose regimens of 3 rPA vaccines and to compare the responses to those following administration of Anthrax Vaccine Adsorbed (AVA or BioThraxTM), the currently available vaccine. The primary immunologic outcome is the proportion of volunteers in each group that mounts an antibody response (defined as a 4-fold or greater increase from pre-vaccination to post-vaccination of anti-rPA IgG antibody with a minimal concentration of 10 µg/ml as measured by ELISA). Secondary outcomes are time to peak response and GMC of anti-PA antibody at peak for each group. In addition, the following immunologic assays will be performed: toxin neutralization assay, oral fluid ELISA, antibody avidity, IgG subclasses, and B-cell memory,T-cell memory and effector subpopulationsThis is a two center study; in which 270 healthy adults aged 18 to 50 years are randomly assigned to 1 of 9 groups; knowledge of rPA product received is double-masked, but schedule and receipt of AVA are unmasked. The duration of study participation is 12 months per volunteer following a screening period of no more than 30 days: administration over a 1- to 4-week period of two doses of IM rPA or 3 doses of SQ AVA with 12-14 follow-up visits. A subset of the approximately 45 volunteers who have agreed to participate in the special immunology subgroup (those with continued antibody responses at 1 year) will be offered extended participation beyond 1 year in which blood is drawn at 18 months, 2 years, 3 years, and 4 years for examination of long-term immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years, inclusive.
2. Good health as evidenced by screening evaluation within the 30 days prior to immunization.
3. Expressed interest and availability to fulfill the study requirements.
4. Signed, informed consents for screening, HIV antibody testing, storing specimens, HIPAA authorization, and protocol-specific research participation.
5. For women of child-bearing potential, agreement to avoid pregnancy for the 30 days following each vaccination by use of highly effective birth control methods. A highly effective birth control method is defined as one which results in a failure rate less than 1% per year when used consistently and correctly. These methods include but may not be limited to the following:

   * Tubal ligation
   * Implantable contraceptive release devices such as Norplant
   * Injected contraceptive hormones such as Depo-Provera
   * Combined oral contraceptives
   * Most IUDs (All commonly used copper and hormone implanted IUDs in the U.S. are highly effective, including the following types: TCu-380A, TCu-220C, MLCu-375, Nova-T, and LNG-20)
   * Vaginal ring hormonal release insertion devices such as NuvaRing
   * Transdermal hormonal contraceptive methods (patches) such as OrthoEvra, and
   * Sexual abstinence
6. Agreement to refrain from taking any experimental drug or vaccine from the day of screening to six months after enrollment.

Exclusion Criteria:

1. History including, but not limited to, any of the following medical illnesses:

   * Diabetes mellitus (not including gestational diabetes that resolved following parturition)
   * Cancer
   * Heart disease, including hospitalization for heart attack or pathologic arrhythmia
   * Unconsciousness, other than concussions or simple faints (vasovagal/syncopal episodes)
   * A seizure disorder (other than simple benign febrile seizures of childhood and petit mal/absence seizures of childhood without manifestations in adulthood)
   * Guillain Barré syndrome
   * Chronic gastrointestinal diseases (including inflammatory bowel disease and celiac disease; not including history of heartburn, gastritis, peptic ulcer disease, or acute gastrointestinal diseases)
   * Recurrent or chronic arthritis, not including overuse injuries or osteoarthritis that does not require daily medication
   * Immunodeficiency
   * Chronic autoimmune diseases, including systemic lupus erythematosus and autoimmune thyroiditis
   * Continuous daily treatment or prophylaxis (other than topical medications) for 6 months duration or more within the last 5 years of a common minor illness such as reactive airway disease, allergic rhinitis/conjunctivitis, or atopic dermatitis (Volunteers with a history of a common minor illness who have required intermittent use of therapeutic or prophylactic medications for less than or equal to 6 months in the last 5 years or for more than 6 months but more than 5 years ago are eligible).
   * Other conditions that in the opinion of the investigator would jeopardize the safety of the subject or the evaluation of the study objectives.
2. Any current illness requiring daily medication (other than vitamins, contraceptives, topical medications, antihistamines, antacids and other reflux medications, smoking cessation medications, headache medications that do not have antipyretic activity, nasal allergy medications, ophthalmologic and otic medications, and thyroxine for stable, inactive hypothyroidism). Volunteers may not take daily oral, nasal, inhaled, or parenteral steroids or non-steroidal anti-inflammatory medications. Medications other than those mentioned above will require approval from the PI, the sponsor, and the medical monitor.
3. Abnormal physical findings including, but not limited to, the following:

   * Cardiac murmur (other than a functional murmur defined as a soft systolic vibratory murmur at the left mid- to lower-sternal border)
   * Focal or global neurologic deficit
   * Hepatomegaly or splenomegaly
   * Lymphadenopathy other than small mobile non-tender nodes in the anterior cervical or inguinal chains or single small nodes in any location
   * Jaundice
   * Hypertension (defined as BP>150/90 on 2 separate days): The blood pressure will be taken by machine or manually at the time of screening and may be repeated once on that day to determine accuracy. If the systolic blood pressure exceeds 150 or diastolic blood pressure exceeds 90, the volunteer will be asked to return another day for a repeat test. If, on repeat, either value is again elevated, the volunteer will be excluded, counseled on appropriate health habits to combat hypertension, and counseled to see his or her doctor.
   * Body Mass Index above 35 or below 18, measured as weight corrected for height (weight in kg/ [height in meters] squared) or weight less than 110 lbs.
   * Other physical findings that in the opinion of the investigator would jeopardize the safety of the subject or the evaluation of the study objectives
4. A current psychiatric condition, including schizophrenia, personality, anxiety, or affective disorders, which in the opinion of the investigator will compromise the subject's ability to participate in the trial
5. Known hypersensitivity to a component of one of the vaccines, including kanamycin (which may be found in trace amounts in rPA[V]) or other aminoglycoside antibiotics, aluminum hydroxide (found in each of the anthrax vaccines), form aldehyde (in AVA), or benzethonium chloride (in AVA).
6. Current drug or alcohol dependence as evidenced by a four-question screening interview to determine whether the subject has had medical, occupational, or family problems related to alcohol or illicit drug use during the past 12 months. These questions are derived from the Drug Abuse Screening Test (DAST 10) developed by the Addiction Research Foundation and recommended by the National Institute for Drug Abuse as a tool for family physicians who wish to routinely screen new patients for drug abuse.
7. History of receipt of anthrax vaccine (licensed or experimental) or history of diagnosis of or exposure to any form of anthrax.
8. Positive serum or urine pregnancy test within the 24 hours prior to each vaccination.
9. Positive blood test for HIV, hepatitis B surface antigen, hepatitis C antibody, or syphilis (defined as positive RPR and FTA).
10. Failure to pass the written exam.
11. Screening laboratory values that fall outside the acceptable study allowable range as delineated in Appendix 1 of the protocol.
12. Receipt of an experimental vaccine or medication within the 30 days prior to enrollment.
13. Receipt of a live, attenuated vaccine within the 30 days prior to enrollment.
14. Receipt of a subunit or killed vaccine within the 14 days prior to enrollment.
15. Receipt of a blood product, including immunoglobulin, in the 90 days prior to enrollment.
16. Donation of a unit of blood within the 56 days prior to enrollment.
17. Anything that, in the opinion of the investigator, will compromise the participation of the volunteer with respect to his/her rights or risks.
18. Oral temperature > 37.7 degrees C or other acute illness occurring prior to inoculation on the day of vaccination. (This circumstance will lead to postponement of enrollment, not exclusion from the trial)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270
Dates: Study Completion 2007-05

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Duke Children's Primary Care, Durham, North Carolina